CLINICAL TRIAL: NCT02096016
Title: Recurrence After Surgery for Cervical Cancer - an Evaluation of the Follow-up Program.
Brief Title: HPV-test, Cervical Cancer and Follow-up
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Follow-up; 1-10-72-323-13
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Human Papilloma Virus; Uterine Cervical Neoplasms; Recurrence
Keywords: Surveillance; Follow up
MeSH Terms: conditions — Uterine Cervical Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Human Papilloma Virus test: Patients treated with surgery alone for uterine cervical neoplasms attending surveillance at Dept. of Obstetrics and Gynecology, Oncogynecological unit, Aarhus University Hospital from 01.01.14 From 01.01.15 patients will be recruited from Oncogynecologic units at Aalborg University Hospital and Rigshospitalet. Recruitment of patients from these institutions has not been successful and has been closed.
  It is expected due to political decisions that the cervical cancer patients from the uptake area of Aalborg University Hospital will be treated at Aarhus University Hospital and they will then be eligible for the study
  Interventions: Procedure: Human Papilloma Virus test from the vaginal vault

INTERVENTIONS:
Procedure: Human Papilloma Virus test from the vaginal vault — Surveillance after surgical treatment of early stage cervical cancer

SUMMARY:
The investigators have planned this project to evaluate the follow-up program after surgery due to cervical cancer and to explore the possibilities for different tests of Human Papilloma Virus (HPV) in contributing to the customization of the follow-up program.

Purpose:

The investigators effort is to provide the background for an evidence-based update of the follow-up program after surgery due to cervical cancer with the purpose of early diagnosis of recurrence affecting quality of life for as few women as possible.

ELIGIBILITY:
Inclusion Criteria:

* Surgery. FIGO stage IA-IB. > 18 years

Exclusion Criteria:

* Ajuvant oncologic treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for cervical cancer.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-01; Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of HPV Genotypes in Vagina (Type 16, 18 and Other) | 2 years

SECONDARY OUTCOMES:
HPV Clearance From Vagina in Between the Two Planned Follow-up Visits. | 2 years

OTHER OUTCOMES:
Evaluate 1-year, 2-year and 5-year Recurrence | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Katrine Fuglsang, MD, Study Director — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes